CLINICAL TRIAL: NCT05480995
Title: Evaluation of Endometriosis With 18F-fluorofuranylnorprogesterone Positron Emission Tomography-Magnetic Resonance Imaging (PET / MRI)
Brief Title: Evaluation of Endometriosis With 18F-fluorofuranylnorprogesterone PET / MRI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-1175; 1P01HD106485-01 (NIH)
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 18F-fluorofuranylnorprogesterone PET / MRI (Experimental): All enrolled subjects will receive the tracer and then have a PET/MRI scan.
  Interventions: Drug: 18F-fluorofuranylnorprogesterone PET / MRI

INTERVENTIONS:
Drug: 18F-fluorofuranylnorprogesterone PET / MRI — Subjects will receive a PET/MRI with 18F-fluorofuranylnorprogesterone tracer

SUMMARY:
Purpose: The aim of this study is to assess the sensitivity and specificity of FFNP PET/MRI for diagnosis of endometriosis.

Participants: A total of 24 participants will be recruited from individuals with clinically suspected endometriosis.

Procedures (methods): This is a prospective, one arm, single center study of 24 subjects with clinically suspected endometriosis to demonstrate FFNP PET-MRI's clinical utility for diagnosis of endometriosis.

ELIGIBILITY:
Inclusion Criteria

* Age 18 or older
* Female of childbearing age (18-55 years)
* Clinically suspected (symptomatic) endometriosis as defined by referring physician (this would also include endometriomas as other disease may be present).
* Scheduled for planned operative laparoscopy with no hormone treatment for at least two cycles
* Able to provide informed consent

Exclusion Criteria

* Male
* Institutionalized subject (prisoner or nursing home patient)
* Known history of breast, ovarian or endometrial cancer.
* Pregnant or breast-feeding women
* Chronic progestin-containing medications or Gonadotropin-releasing hormone (GnRH) analogues in the last 10-16 days (or 2 cycles in the case of GnRH analogues as these are dosed monthly) or inability to discontinue these medications
* Allergy to gadolinium contrast or Glomerular Filtration Rate (GFR) below 30 ml/min.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Subjects must be assigned the gender of female at birth.
Enrollment: 24 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of 18F-fluorofuranylnorprogesterone (FFNP) PET/MR for evaluating endometriosis | Upon completion of all study image data collection for all participants [approximately 1 year]
  The sensitivity of FFNP PET /MR is defined as the ability of readers (radiologists) to correctly detect endometriosis in patients who have endometriosis.
Specificity of 18F-fluorofuranylnorprogesterone (FFNP) PET/MR for evaluating endometriosis | Upon completion of all study image data collection for all participants [approximately 1 year]
  The specificity is similarly defined as the ability of readers to exclude endometriosis in patients who do not have it.

SECONDARY OUTCOMES:
Diagnostic accuracy of PET /MRI | Upon completion of all study image data collection for all participants [approximately 1 year]
  Diagnostic accuracy will be defined by the histologic presence of endometriosis at laparotomy or laparoscopy and/or by symptomatic improvement as defined surgically by the referring physician within 3 months of surgery (surgeon will make final determination).
Correlation of uptake values (SUV-max) with Endometriosis Health Profile (EHP-30) scale controlling for covariates | Upon completion of all study image data collection for all participants [approximately 1 year]
  Diagnostic accuracy will be defined by the histologic presence of endometriosis at laparotomy or laparoscopy and/or by symptomatic improvement as defined surgically by the referring physician within 3 months of surgery (surgeon will make final determination). EHP-30 score is this is the arithmetic mean of 30 questions, each rated 0-100, about function and pain with endometriosis, where 0 indicates the best health status through to 100 worst health status. Scale scores for each scale are calculated from the total of the raw scores of each item in the scale divided by the maximum possible raw score of all the items in the scale, multiplied by 100. The investigators will implement a random effects linear regression model, modeling SUV-max as a function of EHP-30, while controlling for patient-level covariates (BMI, race, age). The investigators will include physician as a random effect to account for physician-level correlation.
Correlation of uptake values (SUV-max) with pain level using a visual analog scale (VAS) controlling for covariates | Upon completion of all study image data collection for all participants [approximately 1 year]
  Diagnostic accuracy will be defined by the histologic presence of endometriosis at laparotomy or laparoscopy and/or by symptomatic improvement as defined surgically by the referring physician within 3 months of surgery (surgeon will make final determination). The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain". The investigators will implement a random effects linear regression model, modeling SUV-max as a function of the pain rating, while controlling for patient-level covariates (BMI, race, age). The investigators will include physician as a random effect to account for physician-level correlation.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Oldan, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina (UNC).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months after and continuing for 36 months following publication
Access Criteria: The investigator who proposes to use the data has approved IRB, IEC, or REB and an executed data use/sharing agreement with UNC.